CLINICAL TRIAL: NCT02441673
Title: Nefopam vs Tramadol in the Prevention of Post Anaesthetic Shivering Following Subarachnoid Block
Brief Title: Nefopam vs Tramadol in the Prevention of Post Anaesthetic Shivering
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lagos State Health Service Commission (Other)
Responsible Party: Principal Investigator, Sarah Beckley, Dr, Lagos State Health Service Commission
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SAS/15/01
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Post Anaesthetic Shivering
Keywords: Postanaesthetic shivering; Subarachnoid block; Tramadol; Nefopam
MeSH Terms: interventions — Nefopam; Tramadol; Metoclopramide; Ranitidine; Meperidine; Ephedrine; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nefopam (Active Comparator): Premedication of IV (Intravenous)10mg Metoclopramide and 50mg Ranitidine would be given morning of surgery to all patients.
  0.15mg/kg of Acupan(Nefopam) would be administered IV after the initiation of the subarachnoid block (Time 0) and presence and severity of shivering (the primary outcome) would be looked out for.
  IV Ephedrine in 3mg alliquots would be given if hypotension occurs; IV oxytocin 30-50mg would be given after delivery of the baby to all patients and IV Pethidine 25mg would be given to abate any residual shivering if a repeat dose of Acupan is not satisfactory.
  Interventions: Drug: Nefopam; Drug: Metoclopramide; Drug: Ranitidine; Drug: Pethidine; Drug: Ephedrine; Drug: oxytocin
- Tramadol (Active Comparator): Premedication of IV (Intravenous)10mg Metoclopramide and 50mg Ranitidine would be given morning of surgery to all patients.
  1mg/kg of tramadol would be administered after the initiation of the subarachnoid block (Time 0) and presence and severity of shivering (the primary outcome) would be looked out for.
  IV Ephedrine in 3mg alliquots would be given if hypotension occurs; IV oxytocin 30-50mg would be given after delivery of the baby to all patients and IV Pethidine 25mg would be given to abate any residual shivering if a repeat dose of Tramadol is not satisfactory.
  Interventions: Drug: Tramadol; Drug: Metoclopramide; Drug: Ranitidine; Drug: Pethidine; Drug: Ephedrine; Drug: oxytocin

INTERVENTIONS:
Drug: Nefopam — Nefopam 0.15mg/kg would be made up to 10mls using sterile water for injection
  Other Names: Acupan
  Arms: Nefopam
Drug: Tramadol — Tramadol 1mg/kg would be made up to 10mls using sterile water for injection
  Arms: Tramadol
Drug: Metoclopramide — 10mg would be given morning of surgery as a prokinetic premedication for all patients.
Drug: Ranitidine — 50mg would be given to each patient morning of surgery as a premedicant to reduce the acidity of the gastric contents. It is routine for CS.
Drug: Pethidine — 25mg would be used to stop shivering where a repeat dose of the primary intervention drugs have not been effective.
Drug: Ephedrine — A vasopressor. Would be used to combat any hypotension that occurs due to the neuroaxial block. Would be used in aliquots of 3mg.
Drug: oxytocin — Would be used for all patients following delivery of the baby to aid contraction of the uterus.

SUMMARY:
Post Anaesthetic Shivering is a common complication of Subarachnoid block. It is graded based on it's severity and has been known to cause various problems like patient's discomfort, hypoxia, change in hemodynamic variables of the patient and poor wound healing. This problem has been managed via pharmacologic and non-pharmacologic means. Non-pharmacologic modalities involve options aimed at warming the patient. Pharmacologically, opioids are used more commonly to prevent and treat this condition. This then introduces the side effect of nausea/vomiting and sedation which may reduce overall patient's satisfaction on the perception of the Subarachnoid block. It is for this reason that Nefopam - a centrally acting non-opioid, non-steroidal anti-inflammatory drug (NSAID) analgesic, relatively new drug in the Nigerian market with significant anti-shivering effect is compared with a well established opioid like Tramadol. Having similar cost profile, the option of replacing Tramadol with Nefopam especially in conditions where the patient is more hemodynamically unstable is considered in this project.

DETAILED DESCRIPTION:
STUDY LOCATION This study would be carried out in Gbagada General Hospital and other General hospitals in Lagos state.

They are all secondary health care facilities with 800 bed spaces in Gbagada and about 3000 in the other centres. Gbagada is a suburban area centrally located in Lagos state and the General hospital was established in 1983.

STUDY DESIGN The study would be a prospective, double-blinded, randomised control study in which both the investigator and the patient would be blinded to the study drugs.

Patients would be randomised into 2 groups. In one group, patients would be given 1mg/kg of tramadol diluted with water for injection to a volume of 10mls. In the second group patients would receive 0.15mg/kg of nefopam diluted with water for injection up to a volume of 10mls.

STUDY POPULATION Patients aged 18 to 45 years with American Society of Anesthesiologists (ASA) physical status II or III scheduled for Caesarean Sessions (CS) amenable to Subarachnoid block who have given written informed consent will be recruited into this study

ANAESTHETIC TECHNIQUE Participants would be randomly divided into 2 groups. Nefopam and Tramadol group via a randomization system.

PREPARATION Patients would be recruited the night before or the morning of surgery. They would be reviewed to allay fear, determine fitness to be part of the study and get consent to join. They would be given the information/consent papers to study and where illiterate or where they do not understand, contents would be explained to them in a language they understand. Verbal and written consent would then be obtained.

After being adequately examined, routine investigations carried out and patient fasted, 2 wide bore Intravenous lines would be sited and the patient weighed. Patients would be routinely given premedication: IV Metoclopramide 10mg and IV Ranitidine 50mg RANDOMIZATION Patient would then be randomly assigned to either of two groups, the tramadol or nefopam group. A randomization schedule would be prepared with sealed envelopes with randomly generated odd and even numbers. The number would be seen only by an assistant who would prepare the chosen medication which are both colourless up to 10mls in an unmarked syringe. Nefopam would be given at 0.15mg/kg and Tramadol 1mg/kg. The patient and Administrator would both be blinded to the content of the syringes. The Assistant with the code would remain within the theatre premises in the event that there is a need to, repeat the chosen drug or break the code in the event of a drug reaction. The theatre environment would be kept at the ambient temperature of between 20 - 25oC and no active warming would be instituted. The Administrator or Researcher would assess each patient for both the primary outcome (shivering) and for the side effects of the study medication.

INDUCTION Baseline vital signs of Non-Invasive Blood Pressure, Mean Arterial Pressure, Pulse Rate, Oxygen Saturation and Temperature measurements would be taken.

Patient would be preloaded with I0mls/kg of Normal saline 15mins before initiation of the block. Placed in the sitting position with a pillow support, routine draping and asepsis would be maintained and using a 25 guage(G) or 26G quincke needle, 12.5mg of 0.5% heavy bupivacaine would be injected at the level of between L2/L3 to L4/L5 interspace. Patient would then be placed supine and given the pre-chosen drug via slow intravenous injection by the assistant who is not part of the study at Time 0 using a Stop Clock.

After the initiation of the block, these parameters would be measured every 5minutes for the first 15mins and every 15 minutes up to 60minutes post initiation of the block. If shivering occurred, the severity would be checked by the principal investigator and a repeat dose of the drug given by the assistant. If this doesn't abate after another 5minutes, a rescue drug of 25mg Pethidine would be given to the patient.

Type of surgery, Bupivacaine dose used, Highest sensory block reached at 10minutes using alcohol swab, Shivering scores, Sedation Scores and Duration of surgery would be documented. Hemodynamic parameters taken at the beginning of surgery would also be recorded every 5minutes for 60minutes.

Hypotension will be defined as less than 20% of the baseline MAP or a value below 60mmHg would be treated by increasing maintenance fluid and Ephedrine using 3mg aliquots.

Incidence of PAS would be determined in both groups; Duration between start of block and onset of PAS and if any other method of stopping PAS was needed to be adopted like repeating the initial dose or IV pethidine 25mg.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients
* Aged 18 to 45 years.
* American Society of Anesthesiologists (ASA) physical status II or III
* Caesarean Sessions (CS) amenable to Subarachnoid block
* Written informed consent

Exclusion Criteria:

* Patients who refuse to sign consent
* Patients with thyroid diseases
* Patients with cardiopulmonary diseases
* Patients with neuromuscular diseases or psychological disorders
* Patients prior on narcotics, sedatives, misoprostol or any medication likely to alter thermoregulation
* Patients with recent history of febrile illness
* Patients with history of malignant hyperthermia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-10-12 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Presence of Post anaesthetic shivering measured by the Crossley and Mahajan Scale | 60 minutes
  Presence of shivering following the subarachnoid block using the Crossley and Mahajan Scale 0 = no shivering
  1. = no visible muscle activity but piloerection, peripheral vasoconstriction or both are present (other causes excluded)
  2. = muscular activity in only one muscle group
  3. = moderate muscular activity in more than one muscle group but no generalized shaking
  4. = muscular activity that involves the whole body
Severity of Post Anaesthetic Shivering measured by th Crossley and Mahajan Scale | 60 minutes
  Severity of shivering where it occurs using the Crossley and Mahajan Scale 0 = no shivering
  1. = no visible muscle activity but piloerection, peripheral vasoconstriction or both are present (other causes excluded)
  2. = muscular activity in only one muscle group
  3. = moderate muscular activity in more than one muscle group but no generalized shaking
  4. = muscular activity that involves the whole body

SECONDARY OUTCOMES:
Presence of Vomiting and Retching using Observation | 60minutes
  Presence or absence of vomiting or retching after administration of the intervention drug
Change in Mean Arterial Pressure (MAP) in mmHg | 60minutes
  Blood Pressure measurement (systolic and diastolic) with the MAP would be measured every 5minutes throughout the 60minutes study duration

CONTACTS AND LOCATIONS:
Overall Officials: Maria Akintimoye, Study Director — Lagos State HealthService Commission